CLINICAL TRIAL: NCT05636163
Title: The Effectiveness of Preoperative Neutrophil-to-lymphocyte and Platelet-to-lymphocyte Ratio in Predicting the Incidence of Nausea and Vomiting After Total Knee Replacement in Hemophilia A
Brief Title: Neutrophil-to-lymphocyte and Platelet-to-lymphocyte Ratio in Predicting the Incidence of Nausea and Vomiting
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, Professor, Qianfoshan Hospital
Other Study IDs: neutrophil-to-lymphocyte ratio
Record Dates: First submitted 2022-11-17; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Hemophilia A
Keywords: Neutrophil; Lymphocyte; Platelet; Hemophilia; Post-operative nausea and vomiting
MeSH Terms: conditions — Hemophilia A; Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
By comparing the incidence of PONV, the dosage of postoperative antiemetic drugs, the postoperative VAS score and the utilization rate of PCIA of hemophilia A patients in the NLR≥2 and NLR<2 groups, investigators could find out the high value in the diagnosis of hemophilia A, which is helpful to guide the clinical diagnosis and treatment of hemophilia A.

DETAILED DESCRIPTION:
Hemophilia arthropathy is a debilitating complication of hemophilia that occurs primarily in severe forms with recurrent spontaneous intra-articular hemorrhage, with the knee being the most commonly affected joint. Currently, total knee arthroplasty is the standard treatment for end-stage hemophilic arthropathy. Due to the special disease of hemophilia, general anesthesia is often chosen as the preferred anesthesia method, and the risk of bleeding is lower than that of neuraxial anesthesia. However, 20 to 30 percent of surgical patients suffer from post-operative nausea and vomiting after general anesthesia. Neutrophil to lymphocyte ratio and platelet to lymphocyte ratio have been suggested as parameters for the diagnosis and follow-up of inflammatory diseases, and inflammation has been found to increase the risk of PONV. However, for patients with hemophilia, no information is currently available on the relationship between the two. In this study, investigators intend to retrospectively analyze the clinical data of patients with hemophilia A in our hospital, explore the clinical value of preoperative NLR and PLR in predicting nausea and vomiting after TKA.

ELIGIBILITY:
Inclusion Criteria:

1. The patients with hemophilia A undergoing unilateral total knee arthroplasty.
2. The age of the patients ranged from 18 to 70 years.
3. American Society of Anesthesiologists is graded as I~III
4. No history of mental illness
5. No history of antiemetic and anticholinergic drugs.
6. No history of serious gastrointestinal diseases.

Exclusion Criteria:

1. Patients who have received long-term steroid treatment
2. Patients who need more than 2.5 mg neostigmine to reverse muscle relaxants
3. Patients with previous malignant tumor, malabsorption, morbid obesity, hypogonadism, thyroid and parathyroid diseases and autoimmune diseases.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemophilia A patients who underwent single knee replacement under general anesthesia in the First Affiliated Hospital of Shandong First Medical University from March 2018 to February 2022
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-01-20 (Estimated); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of PONV in patients with hemophilia A receiving general anesthesia orders for knee arthroplasty | up to 24 hours after surgery
  PONV was defined as the onset of nausea or vomiting within 24 hours after surgery

SECONDARY OUTCOMES:
The amount of postoperative antiemetics | up to 24 hours after surgery
  antiemetics includes ondansetron, metoclopramide, dexamethasone
VAS score after returning to the ward | immediately after returning to the ward
  postoperative pain can be evaluated using the visual analogue scale (0-10 score, 0: no pain, 10: worst imaginable pain).
Usage of PCIA | up to 24 hours after surgery
  the use of postoperative patient controlled intravenous analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Yuelan Wang, Principal Investigator — China, Shandong Qianfoshan Hospital
Locations (1):
- Shandong Provincial Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University, Jinan, Shandong, China